CLINICAL TRIAL: NCT03280563
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating the Efficacy and Safety of Multiple Immunotherapy-Based Treatment Combinations in Patients With Hormone Receptor-Positive HER2-Negative Breast Cancer (MORPHEUS-HR+ Breast Cancer)
Brief Title: A Study of Multiple Immunotherapy-Based Treatment Combinations in Hormone Receptor (HR)-Positive Human Epidermal Growth Factor Receptor 2 (HER2)-Negative Breast Cancer
Acronym: MORPHEUS HR+BC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CO39611; 2017-000335-14 (EudraCT Number)
Record Dates: First submitted 2017-09-11; First posted 2017-09-12 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — atezolizumab; Antibodies; Bevacizumab; entinostat; exemestane; Fulvestrant; ipatasertib; Tamoxifen; abemaciclib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Stage 1: Fulvestrant (Active Comparator): Participants will receive fulvestrant until unacceptable toxicity or disease progression according to RECIST v1.1.
  Interventions: Drug: Fulvestrant
- Stage 1: Atezolizumab + Entinostat (Experimental): Participants will receive doublet combination treatment with atezolizumab plus entinostat until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody; Drug: Entinostat
- Stage 1: Atezolizumab + Fulvestrant (Experimental): Participants will receive doublet combination treatment with atezolizumab plus fulvestrant until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody; Drug: Fulvestrant
- Stage 1: Atezolizumab + Ipatasertib (Experimental): Participants will receive doublet combination treatment with atezolizumab plus ipatasertib until unacceptable toxicity or loss of clinical benefit as determined by the investigator. Prior to enrollment into this arm, the first 6 participants in the study will complete a safety run-in with atezolizumab plus ipatasertib.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody; Drug: Ipatasertib
- Stage 1: Atezolizumab + Ipatasertib + Fulvestrant (Experimental): Participants will receive triplet combination treatment with atezolizumab plus ipatasertib plus fulvestrant until unacceptable toxicity or loss of clinical benefit as determined by the investigator. Prior to enrollment into this arm, the first 6 participants in the study will complete a safety run-in with atezolizumab plus ipatasertib.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody; Drug: Fulvestrant; Drug: Ipatasertib
- Stage 2: Atezolizumab + Bevacizumab + Endocrine Therapy (Experimental): Those who progress or experience unacceptable toxicity during treatment in Stage 1 may be eligible to enter Stage 2. Participants will receive triplet combination therapy with atezolizumab plus bevacizumab plus one of three endocrine therapies (fulvestrant, exemestane, or tamoxifen) selected by the physician. Treatment in Stage 2 will continue until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody; Drug: Bevacizumab; Drug: Exemestane; Drug: Fulvestrant; Drug: Tamoxifen
- Stage 1: Mandatory On-Treatment Biopsy (Experimental): For experimental combination arms that demonstrate clinical activity during the preliminary phase, the Sponsor may open enrollment into a separate mandatory on-treatment biopsy cohort for that combination.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody; Drug: Entinostat; Drug: Fulvestrant; Drug: Ipatasertib; Drug: Abemaciclib
- Stage 1: Atezolizumab + Abemaciclib + Fulvestrant (Experimental): Participants will receive triplet combination treatment with atezolizumab plus abemaciclib plus fulvestrant until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody; Drug: Fulvestrant; Drug: Abemaciclib

INTERVENTIONS:
Drug: Atezolizumab (MPDL3280A), an engineered anti-programmed death-ligand 1 (PD-L1) antibody — Atezolizumab will be given as 840 milligrams (mg) via intravenous (IV) infusion on Days 1 and 15 of each 28-day cycle. This regimen will apply to all arms except when given with entinostat in Stage 1, or exemestane or tamoxifen in Stage 2, in which atezolizumab will be given as 1200 mg via IV infusion on Day 1 of each 21-day cycle.
  Other Names: Tecentriq
  Arms: Stage 1: Atezolizumab + Abemaciclib + Fulvestrant; Stage 1: Atezolizumab + Entinostat; Stage 1: Atezolizumab + Fulvestrant; Stage 1: Atezolizumab + Ipatasertib; Stage 1: Atezolizumab + Ipatasertib + Fulvestrant; Stage 1: Mandatory On-Treatment Biopsy; Stage 2: Atezolizumab + Bevacizumab + Endocrine Therapy
Drug: Bevacizumab — Bevacizumab will be given as 10 milligrams per kilogram (mg/kg) via IV infusion on Days 1 and 15 of each 28-day cycle in the regimen containing fulvestrant. When given with exemestane or tamoxifen, bevacizumab will be given as 15 mg/kg via IV infusion on Day 1 of each 21-day cycle.
  Other Names: Avastin
  Arms: Stage 2: Atezolizumab + Bevacizumab + Endocrine Therapy
Drug: Entinostat — Entinostat will be given as 5 mg orally once a week on Days 1, 8 and 15 of each 21-day cycle.
  Arms: Stage 1: Atezolizumab + Entinostat; Stage 1: Mandatory On-Treatment Biopsy
Drug: Exemestane — Exemestane will be given as 25 mg orally QD in each 21-day cycle.
  Arms: Stage 2: Atezolizumab + Bevacizumab + Endocrine Therapy
Drug: Fulvestrant — Fulvestrant will be given as 500 mg intramuscularly on Days 1 and 15 of Cycle 1 and thereafter on Day 1 of each 28-day cycle.
  Arms: Stage 1: Atezolizumab + Abemaciclib + Fulvestrant; Stage 1: Atezolizumab + Fulvestrant; Stage 1: Atezolizumab + Ipatasertib + Fulvestrant; Stage 1: Fulvestrant; Stage 1: Mandatory On-Treatment Biopsy; Stage 2: Atezolizumab + Bevacizumab + Endocrine Therapy
Drug: Ipatasertib — Ipatasertib will be given as 400 mg orally QD on Days 1-21 of each 28-day cycle.
  Arms: Stage 1: Atezolizumab + Ipatasertib; Stage 1: Atezolizumab + Ipatasertib + Fulvestrant; Stage 1: Mandatory On-Treatment Biopsy
Drug: Tamoxifen — Tamoxifen will be given as 20 mg orally QD in each 21-day cycle.
  Arms: Stage 2: Atezolizumab + Bevacizumab + Endocrine Therapy
Drug: Abemaciclib — Abemaciclib will be given as 150mg twice daily during each 28-day cycle.
  Arms: Stage 1: Atezolizumab + Abemaciclib + Fulvestrant; Stage 1: Mandatory On-Treatment Biopsy

SUMMARY:
This study is designed to evaluate the efficacy, safety, and pharmacokinetics of several immunotherapy-based combination treatments in participants with inoperable locally advanced or metastatic HR-positive, HER2-negative breast cancer who have progressed during or following treatment with a cyclin-dependent kinase (CDK) 4/6 inhibitor in the first- or second-line setting, such as palbociclib, ribociclib, or abemaciclib. The study will be performed in two stages. During Stage 1, participants will be randomized to fulvestrant (control) or an atezolizumab-containing doublet or triplet combination. Those who experience disease progression, loss of clinical benefit, or unacceptable toxicity may be eligible to receive a new triplet combination treatment in Stage 2 until loss of clinical benefit or unacceptable toxicity. New treatment arms may be added and/or existing treatment arms may be closed during the course of the study on the basis of ongoing clinical efficacy and safety as well as the current treatments available.

ELIGIBILITY:
Inclusion Criteria for Both Stages:

* Measurable disease per RECIST v1.1
* Adequate hematologic and end organ function
* Disease progression during or after first- or second-line hormonal therapy with CDK4/6 inhibitor

Inclusion Criteria for Stage 1:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Metastatic or inoperable, locally advanced, histologically or cytologically confirmed invasive HR-positive HER2-negative breast cancer
* Recommended for endocrine therapy, and cytotoxic chemotherapy not indicated at study entry
* Recurrence or progression following most recent systemic breast cancer therapy
* Disease progression during or after first- or second-line hormonal therapy for locally advanced or metastatic disease
* Postmenopausal according to protocol-defined criteria
* Life expectancy >3 months
* Available tumor specimen for determination of PD-L1 status

Inclusion Criteria for Stage 2:

* ECOG performance status of 0-2
* Ability to initiate treatment within 3 months after disease progression or unacceptable toxicity on a Stage 1 regimen

Exclusion Criteria for Both Stages:

* Significant or uncontrolled comorbid disease as specified in the protocol
* Uncontrolled tumor-related pain
* Autoimmune disease except for stable/controlled hypothyroidism, Type 1 diabetes mellitus, or certain dermatologic conditions
* Positive human immunodeficiency virus test
* Active hepatitis B or C
* Active tuberculosis
* Severe infection within 4 weeks and/or antibiotics within 2 weeks prior to study treatment
* Prior allogeneic stem cell or solid organ transplantation
* History of malignancy other than breast cancer within 2 years prior to screening except those with negligible risk of metastasis/death
* History of or known hypersensitivity to study drug or excipients
* For patients entering Stage 2, recovery from all immunotherapy-related adverse events to Grade 1 or better or to baseline at the time of consent

Exclusion Criteria for Stage 1:

* Prior fulvestrant or cytotoxic chemotherapy for metastatic breast cancer, or certain other agents as specified in the protocol
* Unresolved AEs from prior anti-cancer therapy
* Eligibility only for the control arm
* Prior treatment with inhibitors as specified in the protocol

Exclusion Criteria for Stage 2:

* Unacceptable toxicity with atezolizumab during Stage 1
* Uncontrolled cardiovascular disease or coagulation disorder, including use of anticoagulants as specified in the protocol
* Significant abdominal or intestinal manifestations within 6 months prior to treatment
* Grade 2 or higher proteinuria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSF Helen Diller Family CCC, San Francisco, California
  - Stanford Cancer Institute, Stanford, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Wellness Oncology and Hematology - Main Office, West Hills, California
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Providence Cancer Center, Portland, Oregon
  - UPMC Pinnacle Health System, Harrisburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Sch of Med, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
- Israel (5):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- South Korea (3):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - University of Ulsan College of Medicine - Asan Medical Center, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 144 participants with inoperable locally advanced or metastatic hormone receptor-positive (HR+) human epidermal growth factor receptor 2 negative (HER2-) breast cancer took part in the study at 26 investigative sites across the United States of America and South Korea from 22 December 2017 to 26 September 2024. The study is considered "Completed" because all the pre-planned study activities and analyses have been performed.
Pre-assignment Details: The study consisted of two stages: Stage 1: participants were randomized to either the control arm (fulvestrant) or the experimental arms. Stage 2: participants from Stage 1 who experienced unacceptable toxicity, disease progression (PD), or loss of clinical benefit received treatment in Stage 2. Stage 1 participants who did not enter Stage 2 and Stage 2 participants who completed treatment entered the long-term survival follow-up.
Groups:
- Fulvestrant Control: Participants received fulvestrant, 500 milligrams (mg), as an intramuscular (IM) injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter until unacceptable toxicity or PD (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Fulvestrant + Atezolizumab: Participants received fulvestrant (fulv), 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab (atezo) 840 mg as an intravenous (IV) infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Fulvestrant + Atezolizumab + Ipatasertib: Participants received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and ipatasertib (ipat), 400 mg, orally (PO), once a day (QD), on Days 1 to 21 of each 28-day cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Atezolizumab + Ipatasertib: Participants received atezolizumab, 840 mg as an IV infusion on Days 1 and 15 of each cycle along with ipatasertib, 400 mg, PO, QD, on Days 1 to 21 of each 28-day cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Atezolizumab + Entinostat: Participants received atezolizumab, 1200 mg, as an IV infusion on Day 1 of each cycle along with entinostat (entino), 5 mg, PO, once a week on Days 1, 8, and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Fulvestrant + Atezolizumab + Abemaciclib: Participants received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and abemaciclib (abem), 150 mg, PO, twice daily (BID) until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 2: Atezolizumab + Bevacizumab + Fulvestrant: Participants received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and bevacizumab, 10 milligrams per kilogram (mg /kg), as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). Participants who completed Stage 2 treatment entered the long-term survival follow-up.
- Stage 2: Atezolizumab + Bevacizumab + Exemestane: Participants received atezolizumab, 1200 mg, as an IV infusion on Day 1 of each cycle along with bevacizumab, 15 mg/kg, as an IV infusion on Day 1 of each cycle and exemestane, 25 mg, PO, QD during each cycle until unacceptable toxicity, or loss of clinical benefit (1 cycle = 21 days). Participants who completed Stage 2 treatment entered the long-term survival follow-up.
- Stage 2: Atezolizumab + Bevacizumab + Tamoxifen: Participants received atezolizumab, 1200 mg, as an IV infusion on Day 1 of each cycle along with bevacizumab, 15 mg/kg, as an IV infusion on Day 1 of each cycle and tamoxifen, 20 mg, PO, QD during each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days). Participants who completed Stage 2 treatment entered the long-term survival follow-up.
Period: Stage 1
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib | Stage 2: Atezolizumab + Bevacizumab + Fulvestrant | Stage 2: Atezolizumab + Bevacizumab + Exemestane | Stage 2: Atezolizumab + Bevacizumab + Tamoxifen
Started | 25 | 31 | 27 | 6 | 15 | 40 | 0 | 0 | 0
Safety-evaluable (SE) Population (SE population included all participants who received any amount of study treatment.) | 20 | 30 | 26 | 6 | 15 | 39 | 0 | 0 | 0
Completed | 18 | 28 | 24 | 6 | 15 | 33 | 0 | 0 | 0
Not Completed | 7 | 3 | 3 | 0 | 0 | 7 | 0 | 0 | 0
Not completed — Death | 2 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Study Ended by Sponsor | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib | Stage 2: Atezolizumab + Bevacizumab + Fulvestrant | Stage 2: Atezolizumab + Bevacizumab + Exemestane | Stage 2: Atezolizumab + Bevacizumab + Tamoxifen
Started | 0 | 0 | 0 | 0 | 0 | 0 | 13 (6 participants from Stage 1: Atezo+Entino, 3 from Stage 1: Atezo+Ipat, 1 each from Stage 1: Fulv control, Stage 1: Atezo+Fulv, Stage 1: Atezo+Fulv+Ipat and Stage 1: Atezo+Fulv+Abem arms entered this arm in Stage 2.) | 4 (2 participants from Stage 1: Atezo+Fulv+Ipat and 2 participant from Stage 1: Fulv control arms entered this arm in Stage 2.) | 3 (2 participants from Stage 1: Atezo+Fulv and 1 participant from Stage 1: Atezo+Fulv+Ipat arms entered this arm in Stage 2.)
SE Population (SE population included all participants who received any amount of study treatment.) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 4 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Long-term Survival Follow-up
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib | Stage 2: Atezolizumab + Bevacizumab + Fulvestrant | Stage 2: Atezolizumab + Bevacizumab + Exemestane | Stage 2: Atezolizumab + Bevacizumab + Tamoxifen
Started | 15 | 25 | 20 | 3 | 9 | 32 | 11 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 15 | 25 | 20 | 3 | 9 | 32 | 11 | 3 | 3
Not completed — Death | 10 | 14 | 15 | 3 | 6 | 18 | 11 | 1 | 3
Not completed — Study Ended by Sponsor | 4 | 9 | 3 | 0 | 0 | 13 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized population included all participants enrolled, regardless if treatment was received.
Groups:
- Fulvestrant Control: Participants received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter until unacceptable toxicity or PD (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Fulvestrant + Atezolizumab: Participants received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab 840 mg as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Fulvestrant + Atezolizumab + Ipatasertib: Participants received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and ipatasertib, 400 mg, PO, QD, on Days 1 to 21 of each 28-day cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Atezolizumab + Entinostat: Participants received atezolizumab, 1200 mg, as an IV infusion on Day 1 of each cycle along with entinostat, 5 mg, PO, once a week on Days 1, 8, and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Fulvestrant + Atezolizumab + Abemaciclib: Participants received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and abemaciclib, 150 mg, PO, BID until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Total: Total of all reporting groups
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib | Stage 2: Atezolizumab + Bevacizumab + Fulvestrant | Stage 2: Atezolizumab + Bevacizumab + Exemestane | Stage 2: Atezolizumab + Bevacizumab + Tamoxifen | Total
Number analyzed (Participants) | 25 | 31 | 27 | 6 | 15 | 40 | 13 | 4 | 3 | 164
Age, Categorical [Count of Participants; unit: Participants] — Population: Stage 2: The number analyzed is the number of participants who experienced unacceptable toxicity, PD, or loss of clinical benefit in Stage 1 and entered Stage 2 to receive treatment.
  Participants
    Stage 1: number analyzed (Participants) | 25 | 31 | 27 | 6 | 15 | 40 | 0 | 0 | 0 | 144
    Stage 1: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 1: Between 18 and 65 years | 21 | 23 | 22 | 5 | 12 | 28 | 0 | 0 | 0 | 111
    Stage 1: >=65 years | 4 | 8 | 5 | 1 | 3 | 12 | 0 | 0 | 0 | 33
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 4 | 3 | 20
    Stage 2: <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 2: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 3 | 1 | 14
    Stage 2: >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Stage 2: The number analyzed is the number of participants who experienced unacceptable toxicity, PD, or loss of clinical benefit in Stage 1 and entered Stage 2 to receive treatment.
  Participants
    Stage 1: number analyzed (Participants) | 25 | 31 | 27 | 6 | 15 | 40 | 0 | 0 | 0 | 144
    Stage 1: Female | 25 | 31 | 27 | 6 | 15 | 40 | 0 | 0 | 0 | 144
    Stage 1: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 4 | 3 | 20
    Stage 2: Female | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 4 | 3 | 20
    Stage 2: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Stage 2: The number analyzed is the number of participants who experienced unacceptable toxicity, PD, or loss of clinical benefit in Stage 1 and entered Stage 2 to receive treatment.
  Participants
    Stage 1: number analyzed (Participants) | 25 | 31 | 27 | 6 | 15 | 40 | 0 | 0 | 0 | 144
    Stage 1: Hispanic or Latino | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
    Stage 1: Not Hispanic or Latino | 23 | 28 | 25 | 6 | 14 | 40 | 0 | 0 | 0 | 136
    Stage 1: Unknown or Not Reported | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 4 | 3 | 20
    Stage 2: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 2: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 3 | 3 | 19
    Stage 2: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Stage 2: The number analyzed is the number of participants who experienced unacceptable toxicity, PD, or loss of clinical benefit in Stage 1 and entered Stage 2 to receive treatment.
  Participants
    Stage 1: number analyzed (Participants) | 25 | 31 | 27 | 6 | 15 | 40 | 0 | 0 | 0 | 144
    Stage 1: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 1: Asian | 8 | 10 | 11 | 0 | 5 | 15 | 0 | 0 | 0 | 49
    Stage 1: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 1: Black or African American | 1 | 3 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 7
    Stage 1: White | 12 | 16 | 12 | 6 | 9 | 24 | 0 | 0 | 0 | 79
    Stage 1: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 1: Unknown or Not Reported | 4 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 9
    Stage 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 4 | 3 | 20
    Stage 2: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 2: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
    Stage 2: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 2: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 2: White | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 0 | 3 | 15
    Stage 2: More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Stage 2: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Stage 1: Percentage of Participants With Objective Response
Description: Objective response rate (ORR) was defined as the percentage of participants with an objective response of complete response (CR) or partial response (PR) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1). CR was defined as the disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) that have a reduction in short axis to < 10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters (SOD) of all target lesions, taking as reference the baseline SOD, in the absence of CR. Participants with missing or no response assessments were classified as non-responders. Percentages have been rounded off to the nearest whole number.
Time Frame: Up to 50.4 months
Population: Efficacy-evaluable population included all participants who received at least one dose of each drug for their assigned treatment regimen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib
Number analyzed (Participants) | 20 | 30 | 26 | 6 | 15 | 38
percentage of participants | 10.0 [1.23 to 31.70] | 10.0 [2.11 to 26.53] | 26.9 [11.57 to 47.79] | 16.7 [0.42 to 64.12] | 6.7 [0.17 to 31.95] | 26.3 [13.40 to 43.10]
Statistical Analysis 1: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab; Test type: Superiority; Difference in Overall Response Rates = 0.00, 95% CI 2-sided [-21.14 to 21.14]
Statistical Analysis 2: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Ipatasertib; Test type: Superiority; Difference in Overall Response Rates = 16.92, 95% CI 2-sided [-9.03 to 42.88]
Statistical Analysis 3: Comparison: Fulvestrant Control vs Stage 1: Atezolizumab + Ipatasertib; Test type: Superiority; Difference in Overall Response Rates = 6.67, 95% CI 2-sided [-36.76 to 50.09]
Statistical Analysis 4: Comparison: Fulvestrant Control vs Stage 1: Atezolizumab + Entinostat; Test type: Superiority; Difference in Overall Response Rates = -3.33, 95% CI 2-sided [-27.39 to 20.73]
Statistical Analysis 5: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Abemaciclib; Test type: Superiority; Difference in Overall Response Rates = 16.32, 95% CI 2-sided [-6.71 to 39.34]

2. Secondary Outcome: Stage 1: Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to the date of the first recorded occurrence of PD or death from any cause (whichever occurred first) in Stage 1, as determined by the investigator according to RECIST v1.1. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum in the study including baseline in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥ 5 mm. Participants who did not have documented PD or death, PFS was censored at the day of the last tumor assessment. The Kaplan-Meier method was used to estimate the median for PFS.
Time Frame: From randomization to the first occurrence of PD or death (up to 51.9 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib
Number analyzed (Participants) | 20 | 30 | 26 | 6 | 15 | 38
months | 1.95 [1.45 to 4.93] | 3.15 [1.51 to 7.79] | 5.86 [1.64 to 11.24] | 2.28 [1.41 to NA] — The upper limit of the 95% confidence interval (CI) was not estimable due to an insufficient number of participants with events. | 1.82 [1.48 to 3.84] | 6.28 [5.13 to 11.73]
Statistical Analysis 1: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab; Test type: Superiority; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.50 to 1.66]
Statistical Analysis 2: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Ipatasertib; Test type: Superiority; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.35 to 1.20]
Statistical Analysis 3: Comparison: Fulvestrant Control vs Stage 1: Atezolizumab + Ipatasertib; Test type: Superiority; Hazard Ratio (HR) = 1.25, 95% CI 2-sided [0.45 to 3.48]
Statistical Analysis 4: Comparison: Fulvestrant Control vs Stage 1: Atezolizumab + Entinostat; Test type: Superiority; Hazard Ratio (HR) = 1.55, 95% CI 2-sided [0.74 to 3.23]
Statistical Analysis 5: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Abemaciclib; Test type: Superiority; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.28 to 0.88]

3. Secondary Outcome: Stage 1: Clinical Benefit Rate (CBR)
Description: CBR was defined as the percentage of participants with stable disease (SD) ≥ 24 weeks or with confirmed CR or PR, as determined by the investigator according to RECIST v1.1. SD was defined as neither sufficient shrinkage to qualify for CR or PR nor sufficient increase to qualify for PD. CR was defined as the disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) having a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum in the study, including baseline, in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥ 5 mm. Percentages have been rounded off to the nearest whole number.
Time Frame: Up to 51.9 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib
Number analyzed (Participants) | 20 | 30 | 26 | 6 | 15 | 38
percentage of participants | 15.0 [3.21 to 37.89] | 26.7 [12.28 to 45.89] | 42.3 [23.35 to 63.08] | 16.7 [0.42 to 64.12] | 6.7 [0.17 to 31.95] | 42.1 [26.31 to 59.18]

4. Secondary Outcome: Stage 1: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause. Participants who were still alive at the time of OS analysis were censored at the last date they were known to be alive. The Kaplan-Meier method was used to estimate the median for OS.
Time Frame: From randomization to death (up to 62.2 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib
Number analyzed (Participants) | 20 | 30 | 26 | 6 | 15 | 38
months | 26.02 [9.13 to 35.09] | 26.48 [15.87 to 46.46] | 26.91 [20.93 to 47.41] | 10.91 [5.59 to NA] — Upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 23.10 [15.24 to NA] — Upper limit of 95% CI was not estimable due to an insufficient number of participants with events. | 26.71 [22.60 to 36.17]
Statistical Analysis 1: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab; Test type: Superiority; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.36 to 1.65]
Statistical Analysis 2: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Ipatasertib; Test type: Superiority; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.34 to 1.58]
Statistical Analysis 3: Comparison: Fulvestrant Control vs Stage 1: Atezolizumab + Ipatasertib; Test type: Superiority; Hazard Ratio (HR) = 2.26, 95% CI 2-sided [0.55 to 9.34]
Statistical Analysis 4: Comparison: Fulvestrant Control vs Stage 1: Atezolizumab + Entinostat; Test type: Superiority; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.28 to 2.01]
Statistical Analysis 5: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Abemaciclib; Test type: Superiority; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.35 to 1.46]

5. Secondary Outcome: Stage 1: Percentage of Participants Event-free for OS at Month 18
Description: OS was defined as the time from randomization to death from any cause. Participants who were still alive at the time of OS analysis were censored at the last date they were known to be alive. The Kaplan-Meier approach was used to estimate the percentage of participants who were event-free for OS at Month 18. Percentages have been rounded off to the nearest whole number.
Time Frame: At Month 18
Population: Efficacy-evaluable population included all participants who received at least one dose of each drug for their assigned treatment regimen. Overall number analyzed included all participants with data available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib
Number analyzed (Participants) | 10 | 15 | 16 | 6 | 5 | 26
percentage of participants | 63.91 [40.55 to 87.26] | 63.16 [43.97 to 82.35] | 81.61 [65.22 to 98.00] | NA [NA to NA] — The number and 95% CI was not estimable due to an insufficient number of participants with events. | 75.76 [45.17 to 100.00] | 74.40 [59.97 to 88.84]
Statistical Analysis 1: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab; Test type: Superiority; Difference in Event Free Rate = -0.75, 95% CI 2-sided [-30.98 to 29.48]
Statistical Analysis 2: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Ipatasertib; Test type: Superiority; Difference in Event Free Rate = 17.70, 95% CI 2-sided [-10.84 to 46.23]
Statistical Analysis 3: Comparison: Fulvestrant Control vs Stage 1: Atezolizumab + Entinostat; Test type: Superiority; Difference in Event Free Rate = 11.85, 95% CI 2-sided [-26.63 to 50.33]
Statistical Analysis 4: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Abemaciclib; Test type: Superiority; Difference in Event Free Rate = 10.49, 95% CI 2-sided [-16.96 to 37.95]

6. Secondary Outcome: Stage 1: Duration of Response (DOR)
Description: DOR was defined as the time from the first occurrence of a documented objective response (CR or PR) to the first date of recorded PD or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1. CR was defined as the disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) having a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the SOD of all target lesions, taking as reference the baseline SOD, in the absence of CR. PD was defined as at least a 20% increase in the SOD of target lesions, taking as reference the smallest sum in study including baseline in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥ 5 mm. Participants who did not have documented PD or death, DOR was censored at the day of the last tumor assessment. The Kaplan-Meier method was used to estimate the median for DOR.
Time Frame: From first occurrence of a documented OR to the first date of recorded PD or death (up to 50.4 months)
Population: Efficacy-evaluable population included all participants who received at least one dose of each drug for their assigned treatment regimen. Overall number analyzed included participants with an objective response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib
Number analyzed (Participants) | 2 | 3 | 7 | 1 | 1 | 10
months | 13.03 [10.15 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events. | 5.88 [3.29 to NA] — The upper limit of the 95% CI was not estimable due to an insufficient number of participants with events. | 11.07 [7.85 to 20.70] | 4.40 [NA to NA] — The 95% CI was not estimable for a single participant. | 2.46 [NA to NA] — The 95% CI was not estimable for a single participant. | 13.36 [8.87 to 17.02]
Statistical Analysis 1: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab; Test type: Superiority; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.15 to 7.90]
Statistical Analysis 2: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Ipatasertib; Test type: Superiority; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.15 to 4.20]
Statistical Analysis 3: Comparison: Fulvestrant Control vs Stage 1: Fulvestrant + Atezolizumab + Abemaciclib; Test type: Superiority; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.15 to 3.84]

7. Secondary Outcome: Stages 1 and 2: Number of Participants With Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
  SAE = serious adverse events; AESIs = adverse events of special interest.
Time Frame: From baseline until 30 days (for AEs) or 135 days (for SAEs & AESIs) after the last dose of study treatment or until initiation of new systemic anti-cancer therapy, whichever occurred first (Stage 1: up to 52 months; Stage 2: up to 21.7 months)
Population: SE population included all participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib | Stage 2: Atezolizumab + Bevacizumab + Fulvestrant | Stage 2: Atezolizumab + Bevacizumab + Exemestane | Stage 2: Atezolizumab + Bevacizumab + Tamoxifen
Number analyzed (Participants) | 20 | 30 | 26 | 6 | 15 | 39 | 13 | 4 | 3
Participants | 18 | 28 | 26 | 6 | 15 | 39 | 12 | 3 | 3

8. Secondary Outcome: Stage 1: Plasma Concentration of Entinostat
Time Frame: Predose on Day 1 of Cycles 1 and 2; 2-4 hours postdose on Day 1 Cycle 1 (Cycle length = 21 days)
Population: Pharmacokinetic (PK) population included all participants who received at least one dose of atezolizumab and drugs given in combination with atezolizumab during Stage 1. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Stage 1: Atezolizumab + Entinostat
Number analyzed (Participants) | 14
nanograms per milliliter (ng/mL)
  Predose on Cycle 1 Day 1: number analyzed (Participants) | 13
  Predose on Cycle 1 Day 1 | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable as sample were below the limit of quantification (BLQ).
  2-4 Hrs Postdose on Cycle 1 Day 1 | 22.3 (91.0)
  Predose on Cycle 2 Day 1 | 2.12 (60.3)

9. Secondary Outcome: Stage 1: Plasma Concentration of Abemaciclib
Time Frame: Predose on Day 1 of Cycles 1, 2 and 3, and on Day 15 Cycle 1; 4-8 hours postdose on Day 1 Cycle 1 (Cycle length = 28 days)
Population: PK population included all participants who received at least one dose of atezolizumab and drugs given in combination with atezolizumab during Stage 1. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Arm/Group | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib
Number analyzed (Participants) | 31
micrograms per milliliter (µg/mL)
  Predose on Cycle 1 Day 1: number analyzed (Participants) | 3
  Predose on Cycle 1 Day 1 | 0.00417 (50.3)
  4-8 Hour Postdose on Cycle 1 Day 1: number analyzed (Participants) | 25
  4-8 Hour Postdose on Cycle 1 Day 1 | 0.0581 (170.0)
  Predose on Cycle 1 Day 15: number analyzed (Participants) | 30
  Predose on Cycle 1 Day 15 | 0.319 (57.4)
  Predose on Cycle 2 Day 1 | 0.108 (573.7)
  Predose on Cycle 3 Day 1: number analyzed (Participants) | 25
  Predose on Cycle 3 Day 1 | 0.144 (177.7)

10. Secondary Outcome: Stage 1: Plasma Concentration of Ipatasertib
Time Frame: Predose and Postdose at 1 Hour, 2 Hour, 4 Hour, and 6 Hour on Day 15 Cycle 1; Post dose at 1-3 Hour on Day 15 Cycle 3 (Cycle length = 28 days)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Stage 1: Fulv + Atezo + Ipat: Participants received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and ipatasertib, 400 mg, PO, QD, on Days 1 to 21 of each 28-day cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Atezo + Ipat: Participants received atezolizumab, 840 mg as an IV infusion on Days 1 and 15 of each cycle along with ipatasertib, 400 mg, PO, QD, on Days 1 to 21 of each 28-day cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
Arm/Group | Stage 1: Fulv + Atezo + Ipat | Stage 1: Atezo + Ipat
Number analyzed (Participants) | 11 | 2
µg/mL
  Predose on Cycle 1 Day 15 | 0.0353 (248.9) | 0.0105 (10113.9)
  1 Hour Postdose on Cycle 1 Day 15: number analyzed (Participants) | 6 | 2
  1 Hour Postdose on Cycle 1 Day 15 | 0.154 (185.0) | 0.203 (38.5)
  2 Hour Postdose on Cycle 1 Day 15: number analyzed (Participants) | 5 | 1
  2 Hour Postdose on Cycle 1 Day 15 | 0.447 (53.7) | 0.398 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated.
  4 Hour Postdose on Cycle 1 Day 15: number analyzed (Participants) | 5 | 1
  4 Hour Postdose on Cycle 1 Day 15 | 0.273 (45.9) | 0.303 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated.
  6 Hour Postdose on Cycle 1 Day 15: number analyzed (Participants) | 5 | 1
  6 Hour Postdose on Cycle 1 Day 15 | 0.203 (45.4) | 0.227 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated.
  1-3 Hour Postdose on Cycle 3 Day 15: number analyzed (Participants) | 2 | 1
  1-3 Hour Postdose on Cycle 3 Day 15 | 0.576 (25.9) | 0.0664 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated.

11. Secondary Outcome: Stage 1: Plasma Concentration of Fulvestrant
Time Frame: Predose on Day 1 of Cycle 2 and Cycle 3 (Cycle length = 28 days)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Stage 1: Fulv + Atezo + Abem: Participants received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and abemaciclib, 150 mg, PO, BID until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
- Stage 1: Fulve + Atezo: Participants received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab 840 mg as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days). After Stage 1, participants who did not enter Stage 2 entered the long-term survival follow-up.
Arm/Group | Stage 1: Fulv + Atezo + Abem | Stage 1: Fulve + Atezo | Stage 1: Fulv + Atezo + Ipat
Number analyzed (Participants) | 1 | 9 | 7
µg/mL
  Predose on Cycle 2 Day 1 | 0.0127 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 0.0136 (60.2) | 0.0161 (74.3)
  Predose on Cycle 3 Day 1: number analyzed (Participants) | 0 | 6 | 5
  Predose on Cycle 3 Day 1 |  | 0.0107 (40.3) | 0.0121 (38.0)

12. Secondary Outcome: Stage 2: Plasma Concentration of Fulvestrant
Description: Nominal time restarted to 0 at Stage 2. PK data for Stage was analyzed and reported for the subgroups [crossover arms (Stage 1 to Stage 2)] only.
Time Frame: Predose on Day 1 of Cycles 2 and 3 (Cycle length = 21 days)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Stage 1: Atezo + Entino : Stage 2: Atezo + Beva + Fulv: Participants in Stage 1 who received atezolizumab, 1200 mg, as an IV infusion on Day 1 of each cycle along with entinostat, 5 mg, PO, once a week on Days 1, 8, and 15 of each cycle (1 cycle = 21 days), and had PD, entered Stage 2 and received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, and bevacizumab, 10 mg/kg, as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1: Fulv Control : Stage 2: Atezo + Beva+ Fulv: Participants in Stage 1 who received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle (1 cycle = 28 days), and had PD, entered Stage 2 and received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, and bevacizumab, 10 mg/kg, as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1: Atezo + Ipat : Stage 2: Atezo + Beva + Fulv: Participants in Stage 1 who received atezolizumab, 840 mg as an IV infusion on Days 1 and 15 of each cycle along with ipatasertib, 400 mg, PO, QD, on Days 1 to 21 of each cycle (1 cycle = 28 days), and had PD, entered Stage 2 and received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, and bevacizumab, 10 mg/kg, as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
Arm/Group | Stage 1: Atezo + Entino : Stage 2: Atezo + Beva + Fulv | Stage 1: Fulv Control : Stage 2: Atezo + Beva+ Fulv | Stage 1: Atezo + Ipat : Stage 2: Atezo + Beva + Fulv
Number analyzed (Participants) | 3 | 1 | 3
µg/mL
  Predose on Day 1 Cycle 2 (Stage 2) | 0.0207 (14.1) | 0.00938 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 0.0142 (41.2)
  Predose on Day 1 Cycle 3 (Stage 2): number analyzed (Participants) | 2 | 1 | 3
  Predose on Day 1 Cycle 3 (Stage 2) | 0.0121 (39.3) | 0.0175 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 0.0132 (10.3)

13. Secondary Outcome: Stage 2: Serum Concentration of Atezolizumab
Description: Nominal time restarted to 0 at Stage 2; RO5541267 = atezolizumab. PK data for Stage was analyzed and reported for the subgroups [crossover arms (Stage 1 to Stage 2)] only.
Time Frame: Predose on Day 1 of Cycles 1, 2, 3, 4, 8 and 12; 30 minutes (mins) postdose on Day 1 Cycle 1; postdose on Day 120 and Treatment Discontinuation Visit (Cycle length = 21 days)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Groups:
- Stage 1: Fulv + Atezo + Abem : Stage 2: Atezo + Beva + Fulv: Participants in Stage 1 who received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and abemaciclib, 150 mg, PO, BID (1 cycle = 28 days), and had PD, entered Stage 2 and received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, and bevacizumab, 10 mg /kg, as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1: Atezo + Entino : Stage 2: Atezo + Beva + Fulv: Participants in Stage 1 who received atezolizumab, 1200 mg, as an IV infusion on Day 1 of each cycle along with entinostat, 5 mg, PO, once a week on Days 1, 8, and 15 of each cycle (1 cycle = 21 days), and had PD, entered Stage 2 and received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, and bevacizumab, 10 mg /kg, as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1: Fulv + Atezo : Stage 2: Atezo + Beva + Fulv: Participants in Stage 1 who received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab 840 mg as an IV infusion on Days 1 and 15 of each cycle (1 cycle = 28 days), and had PD, entered Stage 2 and received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, and bevacizumab, 10 mg /kg, as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1: Fulv + Atezo : Stage 2: Atezo+ Beva+ Tamo: Participants in Stage 1 who received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then every 4 weeks (Q4W) thereafter along with atezolizumab, 840 mg as an IV infusion on Days 1 and 15 of each cycle (1 cycle = 28 days) and had PD, entered Stage 2 and received atezolizumab, 1200 mg, and bevacizumab, 15 mg/kg, as an IV infusion on Day 1 of each cycle and tamoxifen, 20 mg, PO, QD during each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days).
- Stage 1: Fulv + Atezo + Ipat : Stage 2: Atezo + Beva + Exem: Participants in Stage 1 who received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and ipatasertib, 400 mg, PO, QD, on Days 1 to 21 of each cycle (1 cycle = 28 days), and had PD, entered Stage 2 and received atezolizumab, 1200 mg, and bevacizumab, 15 mg/kg, as an IV infusion on Day 1 of each cycle and exemestane, 25 mg, PO, QD during each cycle until unacceptable toxicity, or loss of clinical benefit (1 cycle = 21 days).
- Stage 1: Fulv + Atezo+ Ipat : Stage 2: Atezo + Beva + Tamo: Participants in Stage 1 who received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, as an IV infusion on Days 1 and 15 of each cycle and ipatasertib, 400 mg, PO, QD, on Days 1 to 21 of each cycle (1 cycle = 28 days), and had PD, entered Stage 2 and received atezolizumab, 1200 mg, and bevacizumab, 15 mg/kg, as an IV infusion on Day 1 of each cycle and tamoxifen, 20 mg, PO, QD during each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 21 days).
- Stage 1: Fulv Control : Stage 2 Atezo + Beva + Exem: Participants in Stage 1 who received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle (1 cycle = 28 days), and had PD, entered Stage 2 and received atezolizumab, 1200 mg, and bevacizumab, 15 mg/kg, as an IV infusion on Day 1 of each cycle and exemestane, 25 mg, PO, QD during each cycle until unacceptable toxicity, or loss of clinical benefit (1 cycle = 21 days).
- Stage 1: Fulv Control : Stage 2: Atezo + Beva+ Fulv: Participants in Stage 1 who received fulvestrant, 500 mg, as an IM injection on Days 1 and 15 of Cycle 1 and then on Day 1 of each cycle (1 cycle = 28 days), and had PD, entered Stage 2 and received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, and bevacizumab, 10 mg /kg, as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
- Stage 1: Atezo + Ipat : Stage 2: Atezo + Beva + Fulv: Participants in Stage 1 who received atezolizumab, 840 mg as an IV infusion on Days 1 and 15 of each cycle along with ipatasertib, 400 mg, PO, QD, on Days 1 to 21 of each cycle (1 cycle = 28 days), and had PD, entered Stage 2 and received fulvestrant, 500 mg, as IM injection on Days 1 and 15 of Cycle 1 and on Day 1 of each cycle thereafter along with atezolizumab, 840 mg, and bevacizumab, 10 mg /kg, as an IV infusion on Days 1 and 15 of each cycle until unacceptable toxicity or loss of clinical benefit (1 cycle = 28 days).
Arm/Group | Stage 1: Fulv + Atezo + Abem : Stage 2: Atezo + Beva + Fulv | Stage 1: Atezo + Entino : Stage 2: Atezo + Beva + Fulv | Stage 1: Fulv + Atezo : Stage 2: Atezo + Beva + Fulv | Stage 1: Fulv + Atezo : Stage 2: Atezo+ Beva+ Tamo | Stage 1: Fulv + Atezo + Ipat : Stage 2: Atezo + Beva + Exem | Stage 1: Fulv + Atezo+ Ipat : Stage 2: Atezo + Beva + Tamo | Stage 1: Fulv Control : Stage 2 Atezo + Beva + Exem | Stage 1: Fulv Control : Stage 2: Atezo + Beva+ Fulv | Stage 1: Atezo + Ipat : Stage 2: Atezo + Beva + Fulv
Number analyzed (Participants) | 1 | 5 | 1 | 2 | 1 | 1 | 1 | 1 | 3
µg/mL
  Predose on Day 1 Cycle 1 (Stage 2): number analyzed (Participants) | 1 | 5 | 1 | 2 | 1 | 1 | 1 | 1 | 2
  Predose on Day 1 Cycle 1 (Stage 2) | 217 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 128 (49.2) | 443 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 160 (209.6) | 277 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 167 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable as samples were BLQ. | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable as samples were BLQ. | 16.3 (63062.7)
  30 mins postdose on Day 1 Cycle 1 (Stage 2): number analyzed (Participants) | 1 | 5 | 1 | 2 | 1 | 1 | 1 | 0 | 2
  30 mins postdose on Day 1 Cycle 1 (Stage 2) | 617 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 388 (22.3) | 907 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 725 (52.9) | 1030 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 679 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 498 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. |  | 491 (16.3)
  Predose on Day 1 Cycle 2 (Stage 2) | 202 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 251 (35.8) | 434 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 211 (143.9) | 373 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 253 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 141 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 136 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 227 (65.2)
  Predose on Day 1 Cycle 3 (Stage 2): number analyzed (Participants) | 0 | 3 | 0 | 2 | 1 | 1 | 0 | 1 | 2
  Predose on Day 1 Cycle 3 (Stage 2) |  | 318 (8.8) |  | 208 (93.2) | 333 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 284 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. |  | 220 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 274 (47.4)
  Predose on Day 1 Cycle 4 (Stage 2): number analyzed (Participants) | 0 | 3 | 0 | 1 | 1 | 1 | 0 | 1 | 2
  Predose on Day 1 Cycle 4 (Stage 2) |  | 302 (20.8) |  | 115 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 341 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 310 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. |  | 238 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 309 (35.2)
  Predose on Day 1 Cycle 8 (Stage 2): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Predose on Day 1 Cycle 8 (Stage 2) |  |  |  |  |  |  |  |  | 131 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated.
  Predose on Day 1 Cycle 12 (Stage 2): number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Predose on Day 1 Cycle 12 (Stage 2) |  |  |  |  |  |  |  |  | 182 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated.
  Postdose on Day 120 (Stage 2): number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1
  Postdose on Day 120 (Stage 2) |  | 27.4 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. |  | 30.0 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. |  |  | 22.6 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. |  | 7.38 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated.
  Treatment Discontinuation Visit (Stage 2): number analyzed (Participants) | 0 | 4 | 1 | 1 | 0 | 0 | 0 | 1 | 3
  Treatment Discontinuation Visit (Stage 2) |  | 250 (18.9) | 450 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 130 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. |  |  |  | 201 (NA) — Since only 1 participant was evaluable, the geometric coefficient of variation could not be estimated. | 169 (145.8)

14. Secondary Outcome: Stage 2: Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab
Description: Participants who received atezolizumab were considered to be treatment-emergent ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following atezolizumab exposure (treatment-induced ADA response), or if they were ADA-positive at baseline and the titer of one or more post-baseline samples was at least 0.60 titer units (t.u.) greater than the titer of the baseline sample (treatment-enhanced ADA response). Participants were considered to be treatment-emergent ADA-negative if they were ADA-negative or were missing data at baseline and all post-baseline samples were negative, or if they were ADA-positive at baseline but did not have any post-baseline samples with a titer that was at least 0.60 t.u. greater than the titer of the baseline sample (treatment unaffected). Participants with a positive post-baseline sample has been reported here.
Time Frame: Post-baseline (up to approximately 134 days)
Population: Pharmacodynamic (PD) population included all participants in the atezolizumab plus entinostat arm with at least one ADA assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: Atezolizumab + Bevacizumab + Fulvestrant | Stage 2: Atezolizumab + Bevacizumab + Exemestane | Stage 2: Atezolizumab + Bevacizumab + Tamoxifen
Number analyzed (Participants) | 10 | 2 | 3
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline until 30 days (for AEs) or 135 days (for SAEs & AESIs) after the last dose of study treatment or until initiation of new systemic anti-cancer therapy, whichever occurred first (Stage 1: up to 52 months; Stage 2: up to 21.7 months) All-cause mortality: Stage 1: up to approximately 62.2 months; Stage 2: From study initiation (from Stage 1) up to approximately 63.7 months)
Description: All-Cause Mortality: Randomized population included all participants enrolled, regardless if treatment was received.
  SAEs and Other AEs: SE population included all participants who received any amount of study treatment.
Arm/Group | Fulvestrant Control | Stage 1: Fulvestrant + Atezolizumab | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Ipatasertib | Stage 1: Atezolizumab + Entinostat | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib | Stage 2: Atezolizumab + Bevacizumab + Fulvestrant | Stage 2: Atezolizumab + Bevacizumab + Exemestane | Stage 2: Atezolizumab + Bevacizumab + Tamoxifen
All-Cause Mortality (participants affected / at risk) | 12/25 | 16/31 | 15/27 | 3/6 | 6/15 | 23/40 | 11/13 | 2/4 | 3/3
Serious Adverse Events (participants affected / at risk) | 2/20 | 3/30 | 12/26 | 3/6 | 4/15 | 14/39 | 1/13 | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 18/20 | 28/30 | 25/26 | 6/6 | 15/15 | 38/39 | 12/13 | 3/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant Control (N=20) | Stage 1: Fulvestrant + Atezolizumab (N=30) | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib (N=26) | Stage 1: Atezolizumab + Ipatasertib (N=6) | Stage 1: Atezolizumab + Entinostat (N=15) | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib (N=39) | Stage 2: Atezolizumab + Bevacizumab + Fulvestrant (N=13) | Stage 2: Atezolizumab + Bevacizumab + Exemestane (N=4) | Stage 2: Atezolizumab + Bevacizumab + Tamoxifen (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myxofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fulvestrant Control (N=20) | Stage 1: Fulvestrant + Atezolizumab (N=30) | Stage 1: Fulvestrant + Atezolizumab + Ipatasertib (N=26) | Stage 1: Atezolizumab + Ipatasertib (N=6) | Stage 1: Atezolizumab + Entinostat (N=15) | Stage 1: Fulvestrant + Atezolizumab + Abemaciclib (N=39) | Stage 2: Atezolizumab + Bevacizumab + Fulvestrant (N=13) | Stage 2: Atezolizumab + Bevacizumab + Exemestane (N=4) | Stage 2: Atezolizumab + Bevacizumab + Tamoxifen (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 4 (8) | 2 (3) | 0 (0) | 1 (1) | 13 (17) | 1 (7) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 10 (26) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 1 (1) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eyelid skin dryness (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 7 (8) | 12 (14) | 3 (3) | 1 (1) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (9) | 14 (33) | 4 (6) | 2 (3) | 33 (55) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 8 (14) | 14 (23) | 4 (6) | 5 (5) | 17 (23) | 5 (5) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (4) | 7 (12) | 3 (4) | 4 (6) | 12 (20) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 11 (13) | 9 (10) | 3 (3) | 4 (4) | 17 (26) | 7 (8) | 1 (1) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 6 (7) | 1 (1) | 3 (4) | 5 (23) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 1 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 4 (5) | 0 (0) | 2 (3) | 6 (13) | 1 (1) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 4 (5) | 0 (0) | 2 (2) | 8 (15) | 2 (2) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 6 (11) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 9 (36) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 5 (11) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wall motion score index abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (8) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 5 (5) | 4 (5) | 4 (4) | 13 (14) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 10 (13) | 3 (4) | 0 (0) | 2 (4) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 2 (3) | 1 (1) | 1 (1) | 10 (12) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 5 (5) | 2 (3) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 4 (5) | 3 (6) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 3 (4) | 2 (4) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 5 (5) | 5 (5) | 0 (0) | 3 (3) | 5 (6) | 3 (6) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (2) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Mood altered (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (9) | 7 (8) | 3 (4) | 4 (4) | 3 (4) | 1 (1) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 9 (12) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 14 (18) | 0 (0) | 1 (1) | 10 (13) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 3 (3) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 6 (8) | 1 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT03280563/Prot_SAP_000.pdf